CLINICAL TRIAL: NCT02293005
Title: Phase II Trial of Alisertib (MLN8237) in Salvage Malignant Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0497; NCI-2014-02568 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-11-11; First posted 2014-11-18 (Estimated); Results first posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Lung Cancer; Mesothelioma
Keywords: Lung Cancer; Mesothelioma; Unresectable malignant pleural mesothelioma; MPM; Alisertib; MLN8237
MeSH Terms: conditions — Lung Neoplasms; Mesothelioma | interventions — MLN 8237

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Alisertib (Experimental): Alisertib administered by mouth at 50 mg twice a day for 7 days in each treatment cycle, followed by a 14-day, treatment-free period.
  Interventions: Drug: Alisertib

INTERVENTIONS:
Drug: Alisertib — 50 mg twice a day on Days 1-7 of each 21-day study cycle.
  Other Names: MLN8237

SUMMARY:
Objectives:

Objectives

The primary objective of this study is to:

To assess 4-month disease control rate (DCR) in pre-treated patients with unresectable malignant pleural mesothelioma (MPM) treated with alisertib

The secondary objectives of this study are to:

To assess the response rate (confirmed and unconfirmed complete + partial responses) To assess the progression-free survival. To assess overall survival. To evaluate the side effects and toxicities associated with this treatment regimen.

To collect archival tissue, blood, pleural effusion fluid and plasma for correlative studies.

Exploratory Objectives:

To collect archival or new tissue, blood and pleural effusion fluid for correlative studies. Tissue biomarkers to be evaluated include aurora kinase pathway and c-myc gene amplification.

Next generation sequencing (NGS) will be conducted on adequate tumor tissue specimens.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will take alisertib tablets by mouth 2 times each day on Days 1-7 of each 21-day study cycle. You must take your doses of alisertib at least 6 hours apart with 1 cup (about 8 ounces) of water.

If you miss or vomit a dose of alisertib, do not retake that dose. Wait and take the next dose as scheduled.

Study Visits:

On Day 1 of Cycles 1-3 and then every odd-numbered cycle after that (Cycles 5, 7, 9 and so on):

* You will have a physical exam.
* Blood (about 4 teaspoons) will be drawn for routine tests.

Every 6 weeks while you are on study, you will have a PET-CT scan of your chest, abdomen, and pelvis to check the status of the disease.

Length of Study:

You may continue taking the study drug for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on this study will be over after you have completed follow-up.

Follow up:

Your study doctor or study team will follow you up 30 days after your last dose by reviewing your medical chart or calling you to see if the side effects are resolved. After that, you will continue to be followed up at 3 months, 6 months and every 6 months beyond that.

The study doctor can explain how the study drug is designed to work.

Up to 58 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
2. Female subject is either: post-menopausal for at least one year before the screening visit, or surgically sterilized, or willing to use an acceptable method of birth control (ie, a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study and at least 1 month after the last dose of alisertib.
3. Male subject, even if surgically sterilized (ie, status postvasectomy), agrees to use an acceptable barrier method for contraception (condom with a spermicidal agent), or completely abstain from heterosexual intercourse during the entire study treatment period through 4 months after the last dose of alisertib.
4. Absolute neutrophil count (ANC) > 1500/mm3, platelets > 100,000/mm3, Hgb > 9 g/dL.
5. Total bilirubin </= 1.5 x upper limit of normal (ULN), SGOT (AST) and SGPT (ALT)< 2.5 x ULN. AST and/or ALT may be up to 5X ULN if with known liver mets
6. Adequate renal function as defined by: Calculated creatinine clearance must be >/= 30 mL/minute
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
8. Pathologic diagnosis of malignant mesothelioma (any primary site is acceptable)
9. Have unresectable malignant mesothelioma (any histology)
10. Received at least one prior pemetrexed-based chemotherapy for unresectable disease, unless within 3 months of receiving platinum-pemetrexed therapy for neoadjuvant or adjuvant treatment that has been unsuccessful.
11. Up to 4 prior lines of systemic therapy (biologic or chemotherapy) are allowed. Maintenance therapy after 4-6 cycles of front-line chemotherapy is still considered 1 line of therapy and is not considered 2 separate therapies.
12. Patients must have measurable disease by modified RECIST or RECIST. Examinations for assessment of measurable disease must have been completed within 28 days prior to registration.
13. Patient must be >/= 18 years of age

Exclusion Criteria:

1. Radiation therapy to more than 25% of the bone marrow. Whole pelvic radiation is considered to be over 25%.
2. Prior allogeneic bone marrow or organ transplantation
3. Known GI disease or GI procedures that could interfere with the oral absorption or tolerance of alisertib. Examples include, but are not limited to partial gastrectomy, history of small intestine surgery with significant removal of the small intestine, and celiac disease
4. Known history of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness, such as severe chronic obstructive pulmonary disease. Patients who use CPAP or BIPAP at night and have controlled sleep apnea syndrome are allowed.
5. Requirement for constant administration of proton pump inhibitor, H2 antagonist, or pancreatic enzymes. Intermittent uses of antacids or H2 antagonists are allowed.
6. Systemic infection requiring IV antibiotic therapy within 14 days preceding the first dose of study drug, or other severe infection.
7. Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
8. Female subject who is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum Beta-human chorionic gonadotropin (Beta-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
9. Patient has received other investigational drugs with 14 days before enrollment
10. Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
11. Other severe acute or chronic medical or psychiatric condition, including uncontrolled diabetes, malabsorption, resection of the pancreas or upper small bowel, requirement for pancreatic enzymes, any condition that would modify small bowel absorption of oral medications, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for enrollment in this study.
12. Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
13. Treatment with clinically significant enzyme inducers, such as the enzyme-inducing antiepileptic drugs phenytoin, carbamazepine or phenobarbital, or rifampin, rifabutin, rifapentine or St. John's wort within 14 days prior to the first dose of alisertib and during the study.
14. Known history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C. Testing is not required in the absence of clinical findings or suspicion. For guidance in defining active infection for hepatitis B, please refer to the WHO guidelines
15. Prior administration of an Aurora A kinase-targeted agent, including alisertib
16. Receipt of corticosteroids within 7 days prior to the first dose of study treatment, unless patient has been taking a continuous dose of no more than 15 mg/day of prednisone for at least 1 month prior to first dose of study treatment. Low dose steroid use for the control of nausea and vomiting will be allowed. Topical steroid use is permitted. Inhaled steroids are permitted.
17. Inability to swallow oral medication or inability or unwillingness to comply with the administration requirements related to alisertib.
18. Administration of myeloid growth factors or platelet transfusion within 14 days prior to the first dose of study treatment.
19. Persons who are incarcerated at time of enrollment (e.g., prisoners) or likely to become incarcerated during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-05-20 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne S. Tsao, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 2015 - February 2017. The patients were recruited in the Thoracic clinic at MD Anderson Cancer Center.
Pre-assignment Details: 28 participants signed consent, 2 participants inevaluable.
Groups:
- Alisertib: Alisertib was administered PO at 50 mg BID for 7 days in each treatment cycle, followed by a 14-day, treatment-free period, for a 21-day cycle.
Period: Overall Study
Arm/Group | Alisertib
Started | 26
Completed | 0
Not Completed | 26
Not completed — Adverse Event | 2
Not completed — Death | 4
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2
Not completed — Progression | 17

BASELINE CHARACTERISTICS:
Arm/Group | Alisertib
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 18
Age, Continuous [Median (Full Range); unit: years] | 69 [44 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 26
Number of Participants with Prior Systemic Therapies [Count of Participants; unit: Participants] | 1

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate at 4 Months
Description: Patients who are free of disease progression at 4 months. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 4 months from treatment started
Population: 1 patient did not complete one cycle of treatment and 25 patients were evaluable for efficacy.
Measure: Count of Participants; unit: Participants
Arm/Group | Alisertib
Number analyzed (Participants) | 25
Participants | 8

2. Secondary Outcome: Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From treatment start, every 6 weeks until progression, death, withdrawal of consent or study completion an average of 25 months
Population: 1 patient did not complete one cycle of treatment and 25 patients were evaluable for efficacy.
Measure: Count of Participants; unit: Participants
Arm/Group | Alisertib
Number analyzed (Participants) | 25
Participants | 1

3. Secondary Outcome: Overall Survival
Description: Overall Survival is defined as the time from the date of randomization to the date of death due to any cause.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 35 months
Population: 1 patient did not complete one cycle of treatment and 25 patients were evaluable for efficacy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alisertib
Number analyzed (Participants) | 25
months | 6.3 [5.7 to 11.1]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of randomization to the date of the first documentation of progressive disease (PD) or date of death, whichever occurs first. Progression is defined using modified Response Evaluation Criteria In Solid Tumors Criteria (mRECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions or RECIST 1.1 if mRECIST cannot be used.
Time Frame: From treatment start to death/progression or last follow-up, whichever come first assessed up to 25 months.
Population: 1 patient did not complete one cycle of treatment and 25 patients were evaluable for efficacy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alisertib
Number analyzed (Participants) | 25
months | 2.8 [1.3 to 4.0]

ADVERSE EVENTS:
Time Frame: Deaths, Serious Adverse Events and Other (Not Including Serious) Adverse events will be captured from the time of the first protocol-specific intervention, until 30 days after the last dose of drug, unless the participant withdraws consent, through study completion an average of 25 months.
Arm/Group | Alisertib
All-Cause Mortality (participants affected / at risk) | 7/26
Serious Adverse Events (participants affected / at risk) | 6/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alisertib (N=26)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alisertib (N=26)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (2)
Allergic reaction (Immune system disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 14 (15)
Anemia (Blood and lymphatic system disorders) | 6 (13)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (2)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Creatinine increased (Investigations) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 11 (12)
Fever (General disorders) | 1 (1)
Gastrointestinal disorders - (Other), specify (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions - (Other), specify (General disorders) | 3 (6)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 7 (9)
Musculoskeletal and connective tissue disorder - Specify (Other) (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (10)
Neutrophil count decreased (Investigations) | 3 (5)
Non-cardiac chest pain (General disorders) | 1 (2)
Oral pain (Gastrointestinal disorders) | 2 (2)
Platelet count decreased (Investigations) | 5 (7)
Reproductive system and breast disorders - (Other), specify (Reproductive system and breast disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin and subcutaneous tissue disorders - (Other), specify (Skin and subcutaneous tissue disorders) | 2 (2)
Somnolence (Nervous system disorders) | 4 (5)
Thromboembolic event (Vascular disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (7)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT02293005/Prot_SAP_000.pdf